CLINICAL TRIAL: NCT06553144
Title: Comparative Analysis of Intra-canal Photodynamic Therapy With Different Photosensitizers on Periapical Healing
Brief Title: Comparative Analysis of Photodynamic Therapy on Periapical Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Reyhan Ece Ari, lecturer, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gaziantep Ünivesitesi 2019/259
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Methylene Blue; Erythrosine; Curcumin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Curcumin (Experimental): patient with single root and canal, along with apical radiolucent lesions
  Interventions: Procedure: curcumin
- Erythrosine B (Experimental): patient with single root and canal, along with apical radiolucent lesions
  Interventions: Procedure: erythrosine b
- Control (Active Comparator): patient with single root and canal, along with apical radiolucent lesions
  Interventions: Procedure: control
- Methylene Blue (Experimental): patient with single root and canal, along with apical radiolucent lesions
  Interventions: Procedure: methylene blue

INTERVENTIONS:
Procedure: control — Canals were irrigated with only10 mL of 5% NaOCl
  Arms: Control
Procedure: methylene blue — 0.1 mg/mL methylene blue solition delivered into the canal and irradiated with a 100mW diode laser at a wavelength of 660 nm
  Arms: Methylene Blue
Procedure: erythrosine b — 0.3 mg/mL eryrhtosine b solition delivered into the canal and irradiated with a 100mW diode laser at a wavelength of 660 nm
  Arms: Erythrosine B
Procedure: curcumin — 5.0 mg/mL curcumin solition delivered into the canal and irradiated with a 200mW diode laser at a wavelength of 450 nm
  Arms: Curcumin

SUMMARY:
As a result of tooth decay, lesions caused by infection occur at the root tip. These teeth can heal with root canal treatment. In this study, additional applications will be made to increase the success of root canal treatment. The materials we will use are harmless. At the end of the procedure, your teeth will be monitored regularly and their healing status will be checked.

DETAILED DESCRIPTION:
Root canal therapy seeks to eradicate root canal infections and prevent their recurrence. Given the intricate nature of the root canal system and biofilm formations, achieving complete disinfection with current techniques is challenging. Nevertheless, it has been noted that residual microorganisms within the root canal contribute significantly to either the healing or the development of apical periodontitis. Various methods, such as sonic and ultrasonic activation, laser application, and PDT (Photodynamic Therapy), have been proposed in literature to enhance root canal disinfection.

Several in vivo and in vitro studies have demonstrated a significant reduction in bacterial load following PDT adjunct to root canal therapy. However, long-term in vivo outcomes of PDT as a complement to root canal disinfection remain scarce. From an endodontic perspective, many photosensitizers have not undergone clinical evaluation. This study seeks to assess the impact of PDT using different photosensitizers on in vivo lesion healing.

First of all, teeth that met the inclusion criteria were planned to be randomly divided into 4 groups. However, in this case, gender and tooth numbers would not be distributed equally among the groups. Therefore, a stratified randomization method was employed to ensure balanced distribution of participants across the four study groups based on gender (male, female) and tooth type (anterior, premolar). To ensure an unbiased distribution of teeth across four treatment groups (Curcumin, Methylene Blue, Erythrosine B, and Control) a randomization process was implemented using Excel VBA (Visual Basic for Applications) by a third party not involved in the study intervention.

Vitality tests yielded negative results for all teeth. The treatments were administered consistently by the same operator to ensure uniformity. However, due to irregular attendance at follow-up appointments by six patients and one instance of tooth extraction, the study ultimately involved 70 teeth, as elaborated in. , Study Design Participants were randomized into four groups. Periapical radiographs of the teeth were captured using a dental X-ray unit (Satalect X-Mind, France) set at 250 kV, 4 mA, and 0.12 seconds of irradiation time, employing a parallel technique guided by a cone indicator. For teeth with indistinct lesion sizes on periapical radiographs, three-dimensional images were acquired using cone beam computed tomography (CBCT) (Planmeca, Helsinki, Finland) with settings of 90 kVp, 12 mA, 14 seconds, and a 16x5 imaging field.

Following rubber dam isolation, access cavities were prepared using a diamond bur. The working length was determined using a 15 K-file (Dentsply Maillefer, Ballaigues, Switzerland) coupled with an apex locator (Root ZX, Morita, Japan), ensuring a 0.5 mm short of the "00" point. Radiographic confirmation of the working length was obtained.

Canal instrumentation up to a 20 K-file was carried out, followed by further preparation using the R25 Reciproc instrument (VDW, Munich, Germany) operated by a VDW Silver endodontic motor (VDW) at the Reciproc All setting. After three pecking motions, irrigation with 5% Sodium hypochlorite (NaOCl) (Werax, İzmir, Türkiye) was conducted until the full canal length was reached. Mechanical instrumentation is completed with the R40 instrument.

Throughout the procedure, each canal received irrigation with 10 mL of 5% NaOCl at a flow rate of 0.1 ml/sec via a 30-G irrigation needle (Endo-Top Wola, Poland), positioned 1 mm short of the working length. Subsequently, canals were rinsed with distilled water and then irrigated with 5 mL of 17% EDTA (Kemiger, Ankara, Turkey) for 1 minute, allowing an additional 1-minute dwell time. Ultrasonic activation involved using 2 mL of NaOCl in total, administered three times for 20 seconds each, employing a Niti U-File #25 attached to the E2 tip of an ultrasonic device (Woodpecker, China) in endodontic mode, positioned 1 mm short of the working length. After each irrigation step, canals were rinsed with distilled water.

Following this stage, participants were allocated into four groups for the final irrigation protocol. The randomization process determined which protocol would be performed for each tooth and was performed by a blinded assistant.

Group 1: A curcumin solution was prepared by dissolving curcumin (Sigma-Aldrich, Steinheim, Germany) in 0.5% dimethyl sulfoxide (DMSO) (Aromel Medikal, Konya, Türkiye) to achieve a final concentration of 5.0 mg/mL. The photosensitizer was delivered into the canal using an irrigation needle until the pulp chamber was filled. After a 3-minute wait, ultrasonic activation was performed for 20 seconds. The solution was then refreshed, and the activation process was repeated two more times for a total of 60 seconds. The last refreshed photosensitizer was irradiated with a 200mW diode laser (SiroLaser Blue, Dentsply, Germany) at a wavelength of 450 nm, employing spiral movements with an EasyTip 200 µm Endo fiber optic tip for 20 seconds. This process was repeated two more times. Finally, the photosensitizer was rinsed with distilled water.

Group 2: Erythrosine B (Sigma Aldrich, St. Louis, MO, USA) was diluted with phosphate-buffered saline solution to achieve a final concentration of 0.3 mg/mL. Ultrasonic activation was performed similarly to Group 1, but laser application utilized a wavelength of 660 nm and a power of 100 mW.

Group 3: Methylene blue (Sigma-Aldrich, Germany) at a concentration of 0.1 mg/mL was introduced into the canal as in the previous groups and activated by both ultrasonic and laser methods. The parameters for this group were also set to a wavelength of 660 nm and a power of 100 mW.

Group 4: Canals were irrigated with 10 mL of 5% NaOCl at a flow rate of 0.1 mL/sec.

All canals were subsequently rinsed with distilled water. The final irrigation involved the use of 2 mL of 1% EDTA for 1 minute. A 40/04 master gutta-percha cone was placed and confirmed radiographically. Canals were dried using sterile paper points. The obturation of canals with the 40/04 gutta-percha cones was carried out using Endoplus (President/München/ Germany) and the lateral condensation technique. Following the removal of excess gutta-percha, access cavities were cleaned with alcohol and restored incrementally with resin-modified glass ionomer cement (Riva Light Cure HV, Australia) and composite resin (G-Premio Bond, Tokyo, Japan).

Participants were scheduled for follow-up appointments at 6, 12, and 24 hours, as well as at 1 week, during which they were asked to report any pain experienced. Pain levels were assessed using the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (most severe pain), and recorded accordingly. Subsequent follow-up appointments were scheduled at 1, 3, 6, and 9 months, and a final 1-year follow-up, during which radiographs were taken to monitor the healing of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Encompassed lower premolars
* Upper central and lateral incisors with a single root and canal, along with apical radiolucent lesions

Exclusion Criteria:

* Periodontal pockets exceeding 4 mm,
* Mobility,
* Nonrestorability,
* Immaturity,
* any indications of fracture or dental anomalies
* chronic drug users

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
healing of periapical lesions by radiography | long-term follow-up evaluation in 12 months
  The area of lesions in periapical radiographs, captured using the parallel technique, was calculated in mm² utilizing Image J 1.28 software (Figure 7) (National Institute of Health, USA).
post-op pain | Participants were scheduled for follow-up appointments at 6, 12, and 24 hours, as well as at 1 week,
  Participants were scheduled for follow-up appointments at 6, 12, and 24 hours, as well as at 1 week, during which they were asked to report any pain experienced. Pain levels were assessed using the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (most severe pain), and recorded accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: REYHAN ECE ARI, Study Director — University of Gaziantep
Locations (1):
- Gaziantep Üniversitesi, Gaziantep, Adana, Turkey (Türkiye)